CLINICAL TRIAL: NCT05823948
Title: A Study to Evaluate Flash Glucose Monitoring Based Titration of Once-weekly Insulin Icodec in Insulin-naïve Participants With Type 2 Diabetes
Brief Title: A Study Using Flash Glucose Measurements for a New Once-weekly Insulin (Insulin Icodec) in People With Type 2 Diabetes Who Have Not Used Insulin Before (ONWARDS 9)
Acronym: ONWARDS 9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4909; U1111-1271-9296 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Insulin Icodec (Experimental): Participants will receive 70 Units (U) insulin icodec subcutaneously once-weekly for 26 weeks.
  Interventions: Drug: Insulin Icodec

INTERVENTIONS:
Drug: Insulin Icodec — Participants will receive insulin icodec once-weekly subcutaneously into the thigh, upper arm or abdomen.

SUMMARY:
This study looks at how a person with type 2 diabetes can be treated with insulin icodec and a flash glucose monitor (a small sensor inserted under the skin to measure blood sugar all the time). The study will look at how well insulin icodec controls blood sugar when used in combination with a flash glucose monitor. Participants will get insulin icodec that they have to inject once a week on the same day of the week. The insulin will be injected with a needle in a skin fold in the thigh, upper arm, or stomach. The study will last for about 8 months. Participants will have to wear a flash glucose monitor throughout the study. This is a sensor that fits on arm. Participants will be asked to use a commercially available app called LibreView to allow team to view flash glucose monitor data. Participants will get a study phone to scan the flash glucose monitor 4 times daily and they will be able to see all of the flash glucose monitor data during the study. Women cannot take part if pregnant, breast-feeding or planning to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study
* Age above or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes (T2D) greater than or equal to (>=) 180 days before screening
* HbA1c from 7.0%-11.0% (53.0-96.7 millimoles per mole [mmol/mol]) both inclusive at screening confirmed by central laboratory analysis
* Insulin-naïve. However, short term insulin treatment for a maximum of 14 consecutive days before screening is allowed, as is prior insulin treatment for gestational diabetes
* Stable daily dose(s) >=90 days before screening of any of the following antidiabetic drug(s) or combination regimen(s) at effective or maximum tolerated dose as judged by the investigator:

  1. Any metformin formulations >= 1500 milligrams (mg) or maximum tolerated or effective dose or
  2. Any metformin combination formulations >=1500 mg or maximum tolerated or effective dose or
  3. Other antidiabetic Drugs including combination products (>=half of the maximum approved dose according to local label or maximum tolerated or effective dose) of the classes specified below: Sulfonylureas, Meglitinides (glinides), Dipeptidyl peptidase-4 (DPP-4) inhibitors, Sodium-dependent glucose cotransporter 2 (SGLT2) inhibitors, Thiazolidinedione, Alpha-glucosidase inhibitors, Oral combination products (for the allowed individual oral antidiabetic drugs, Oral or injectable glucagon-like peptide-1 (GLP-1) receptor agonists
* Intensification with basal insulin is indicated to achieve fasting glycaemic target (4.4-7.2 millimoles per liter [mmol/L]; 80-130 milligrams per deciliter [mg/dL]) at the discretion of the treating investigator
* Body mass index (BMI) less than or equal to (<=) 40.0 kilograms per meter square (kg/m^2)

Exclusion Criteria:

* Unwilling or unable to avoid concomitant medication e.g., ascorbic acid (vitamin C) that can influence the flash glucose monitoring (FGM) sensor throughout the study and contraindications e.g., implanted medical devices such as pacemakers
* Any episodes of diabetic ketoacidosis within 90 days before screening as declared by the participant or in the medical records
* Myocardial infarction, stroke, transient ischaemic attack or hospitalisation for unstable angina pectoris within 180 days before the day of screening and between screening and initiation visits
* Chronic heart failure classified as being in New York Heart Association (NYHA) Class IV at screening
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g., treatment with orlistat, thyroid hormones, or corticosteroids)
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before the day of screening or in the period between screening and initiation visits. Pharmacological pupil dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From initiation week 0 (Visit 3) to week 26 (Visit 26)
  Measured in percentage (%)-point.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (20):
- United States (20):
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Clinical Trials Research_Sacramento_0, Sacramento, California
  - San Diego Family Care, San Diego, California
  - Mills-Peninsula Hlth Services, San Mateo, California
  - Florida Inst For Clin Res LLC, Orlando, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - East West Med Res Inst, Honolulu, Hawaii
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Accellacare_NC, Wilmington, North Carolina
  - Diabetes & Endocrinology Asso, Canton, Ohio
  - AM Diabetes And Endocrinology, Bartlett, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - Velocity Clin Res, Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Fmc Science, Llc, Lampasas, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, San Antonio, Texas
  - Chrysalis Clinical Research, St. George, Utah

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Bergenstal RM, Asbjornsdottir B, Johanning Bari T, Hulkund S, Winhofer Y, Wysham C. Continuous Glucose Monitoring-Based Titration of Once-Weekly Insulin Icodec in Insulin-Naive Individuals with Type 2 Diabetes (ONWARDS 9): A Phase 3b, Multicenter, Single-Arm, Treat-to-Target Clinical Trial. Diabetes Technol Ther. 2025 Jul;27(7):527-536. doi: 10.1089/dia.2025.0050. Epub 2025 Mar 5. PMID 40040516